CLINICAL TRIAL: NCT03141060
Title: A Phase I/II Open-Label, Single-Arm Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Delamanid in Combination With Optimized Multidrug Background Regimen (OBR) for Multidrug-Resistant Tuberculosis (MDR-TB) in Children With MDR-TB With and Without HIV
Brief Title: Evaluating the Pharmacokinetics, Safety, and Tolerability of Delamanid in Combination With Optimized Multidrug Background Regimen (OBR) for Multidrug-Resistant Tuberculosis (MDR-TB) in HIV-Infected and HIV-Uninfected Children With MDR-TB
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMPAACT 2005; 20721 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2017-05-01; First posted 2017-05-04 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Tuberculosis; HIV Infections
MeSH Terms: conditions — Tuberculosis; HIV Infections | interventions — OPC-67683

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1: Delamanid (Experimental): Participants will receive delamanid (DLM) twice daily for 24 weeks. Participants will also receive non-study prescribed OBR for MDR-TB.
  Interventions: Drug: Delamanid; Drug: Optimized multidrug background regimen (OBR) for children with MDR-TB

INTERVENTIONS:
Drug: Delamanid — Administered orally; dosing will be based on participants' age and weight.
  Other Names: DLM
Drug: Optimized multidrug background regimen (OBR) for children with MDR-TB — Non-study prescribed OBR will vary according to local, national, and/or international guidelines for treatment of children with MDR-TB. Administered in addition to DLM for 24 weeks.

SUMMARY:
This study will evaluate the pharmacokinetics, safety, and tolerability of the anti-tuberculosis (TB) drug delamanid (DLM) in combination with an optimized multidrug background regimen (OBR) for multidrug-resistant tuberculosis (MDR-TB) in HIV-infected and HIV-uninfected children with MDR-TB.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the pharmacokinetics, safety, and tolerability of the anti-TB drug DLM in combination with OBR for MDR-TB in HIV-infected and HIV-uninfected children with MDR-TB.

Participants will be enrolled in one of four age cohorts: 12 to less than 18 years, 6 to less than 12 years, 3 to less than 6 years, or 0 to less than 3 years. All participants will receive DLM dosed according to their age group and weight for 24 weeks.

Study visits will occur at study entry; Weeks 2 and 4; every 4 weeks through Week 40; and at Weeks 48, 60, 72, and 96. Visits may include physical examinations; blood, urine, and sputum collection; chest x-rays; electrocardiograms (ECGs); hearing tests; adherence assessments; and acceptability questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Parent (or legal guardian) is willing and able to provide written informed consent for child study participation. Additionally, for children whose assent is required per site institutional review board/ethics committee (IRB/EC) policies and procedures, child is willing and able to provide written assent for his or her study participation.
* Age less than 18 years at enrollment
* HIV-uninfected, or HIV-infected (see the protocol for more information on this criterion)
* If HIV-infected: Initiated the standard of care antiretroviral therapy (ART) regimen at least two weeks prior to enrollment (note: regimens including efavirenz [EFV], nevirapine [NVP], a boosted protease inhibitor [PI], or integrase strand transfer inhibitor [INSTI] are allowed)
* Confirmed or probable MDR-TB classified as follows:

  * Confirmed MDR-TB (or rifampicin mono-resistant TB [RMR-TB], pre-extensively drug-resistant [XDR] or XDR-TB):

    * Intra-thoracic (pulmonary) TB based on chest radiograph consistent with TB, and/or any of the following forms of extrathoracic TB:
    * 1) Peripheral TB lymphadenitis
    * 2) Pleural effusion or fibrotic pleural lesions
    * 3) Stage 1 TB meningitis
    * 4) Miliary and abdominal TB
    * 5) Other non-disseminated forms of TB disease (see also exclusion criterion below)
    * AND
    * Microbiological confirmation of Mycobacterium tuberculosis from any clinical specimen by either culture or molecular methods (including Xpert MTB/RIF)
    * AND
    * Drug-resistance demonstrated by genotypic (molecular) or phenotypic methods, with any of the following resistance patterns:
    * MDR-TB (resistance to both rifampicin and isoniazid)
    * RMR-TB or where additional isoniazid (INH) resistance has not been confirmed (i.e., isolated Xpert MTB/RIF rifampicin resistance)
    * Pre-XDR-TB (MDR-TB plus resistance to either a fluoroquinolone or a second-line injectable agent)
    * XDR-TB (MDR-TB plus resistance to both a fluoroquinolone and a second-line injectable)
    * Note: RMR-TB, MDR-TB, pre-XDR-TB and XDR-TB are therefore collectively referred to as "MDR-TB" for the purposes of the protocol
  * Probable MDR-TB (or RMR, pre-XDR or XDR-TB), with inclusion of intrathoracic and/or extrathoracic TB as listed below:

    * A presumptive diagnosis of intrathoracic (pulmonary) TB based on well-documented clinical symptoms or signs of TB AND chest radiograph consistent with TB, and/or any of the following forms of extrathoracic TB:
    * Peripheral TB lymphadenitis
    * Pleural effusion or fibrotic pleural lesions
    * Stage 1 TB meningitis
    * Miliary and abdominal TB,
    * Other non-disseminated forms of TB disease (see also exclusion criterion below)
    * AND
    * One of the following:
    * Exposure to a confirmed MDR-TB source case* (RMR-TB, pre-XDR-TB, XDR-TB)
    * Documented failure to respond to a first-line regimen, and where adherence was well documented.
    * AND
    * The clinical decision has been made to treat for MDR-TB
    * * Confirmed MDR-TB source cases defined as a case with intrathoracic TB with or without extrathoracic TB, with microbiological confirmation of Mycobacterium tuberculosis from any clinical specimen by either culture or molecular methods (including Xpert MTB/RIF), and with drug-resistance demonstrated by genotypic (molecular) or phenotypic methods, with any of the resistance patterns described above.
* Albumin level greater than 2.8 g/dL within 30 days prior to enrollment
* Potassium greater than 3.4 and less than 5.6 mmol/L; magnesium greater than 0.59 mmol/L within 30 days prior to enrollment. Note: Electrolytes can be repleted and a recheck may be performed to meet eligibility criteria.
* BMI Z-score greater than -3 for children greater than or equal to 5 years of age; weight for length/height Z-score greater than -3 for children less than 5 years of age (using latest World Health Organization scores), at screening
* Weight greater than or equal to 3 kg, at screening
* Has initiated an appropriate optimized background regimen (OBR) MDR-TB treatment regimen as per routine treatment decision, at least two weeks but not more than eight weeks prior to enrollment, and in the opinion of the site investigator, is tolerating the regimen well at enrollment. Note: An appropriate OBR MDR-TB treatment regimen is defined as including components based on the sensitivities of the infecting isolate, if known, and past treatment history, if known. This regimen should also follow the OBR MBR-TB treatment guidelines as described in the protocol.
* If male and engaging in sexual activity that could lead to pregnancy of the female partner: Agrees to use a barrier method of contraception (i.e. male condom) throughout the first 28 weeks on study (i.e., until four weeks after discontinuation of DLM).
* If female and of reproductive potential, defined as having reached menarche and not having undergone a documented sterilization procedure (hysterectomy, bilateral oophorectomy, or salpingectomy): Negative pregnancy test at screening within 14 days prior to enrollment.
* If female, of reproductive potential (as defined in the protocol), and engaging in sexual activity that could lead to pregnancy: Agrees to avoid pregnancy and to use one of the following forms of birth control while receiving DLM and for one month after stopping DLM: condoms, diaphragm or cervical cap, intrauterine device (IUD), hormonal-based contraception. The selected method must be initiated prior to enrollment.

Exclusion Criteria:

* Known allergy to any nitroimidazoles or nitroimidazole derivatives
* Active use of prohibited medications listed in the protocol, within 3 days of enrollment
* Participant has a history of any of the following, as determined by the site investigator or designee based on maternal report and available medical records:

  * A significant cardiac arrhythmia that requires medication or a history of heart disease (heart failure, coronary artery disease) that increases the risk for Torsade de Pointes
  * Significant gastrointestinal (GI), metabolic, neuropsychiatric, kidney or endocrine disease at screening that would, in the investigator's opinion, preclude safe participation in the trial and/or assessment of primary endpoints
  * Previous DLM or pretomanid exposure
  * Note: Participants can have received up to 14 + 3 days (i.e., up to 17 days) of DLM prior to enrollment
* Abnormal electrocardiogram (ECG) (including QTcF [mean value of QT interval, corrected using Fredericia correction, on ECG performed in triplicate] greater than or equal to 450 ms, atrioventricular block, or prolonged QRS greater than or equal to 120 ms) at screening
* Karnofsky score less than 30% for participants greater than or equal to 16 years of age or Lansky play score less than 30% for participants less than 16 years of age, at screening
* Alcohol intake that in the opinion of the study investigator could potentially interfere with study participation and/or introduce safety concerns with use of DLM
* Lactating with plans to breastfeed, at enrollment
* Tuberculous meningitis (TBM) Stage 2 or 3, or osteo-articular TB at screening
* Co-enrolled in any other trial involving pharmacologic regimens, at screening
* If HIV-exposed and less than 2 years of age: Breastfeeding at enrollment

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2025-04-22 (Actual); Study Completion 2025-05-29 (Actual)

PRIMARY OUTCOMES:
Frequency of Grade 3 or 4 adverse events (AEs) | Measured through Week 24
  Based on labs, signs/symptoms, diagnoses
Frequency of Grade 3 or 4 AEs judged by the Clinical Management Committee (CMC) to be related to DLM | Measured through Week 24
  Based on labs, signs/symptoms, diagnoses
Frequency of permanent discontinuations of DLM due to a toxicity or AE | Measured through Week 24
  Based on study drug discontinuation criteria outlined in the protocol
Frequency of QTcF interval greater than or equal to 500 ms | Measured through Week 24
  Based on electrocardiogram (ECG)
Frequency of participant deaths | Measured through Week 24
  Grade 5 event

SECONDARY OUTCOMES:
Frequency of Grade 3 or 4 AEs | Measured through Week 72
  Based on labs, signs/symptoms, diagnoses
Frequency of Grade 3 or 4 AEs judged by the CMC to be related to DLM | Measured through Week 72
  Based on labs, signs/symptoms, diagnoses
Frequency of permanent discontinuations of DLM due to a toxicity or AE | Measured through Week 72
  Based on study drug discontinuation criteria outlined in the protocol
Frequency of QTcF interval greater than or equal to 500 ms | Measured through Week 72
  Based on ECG
Frequency of participant deaths | Measured through Week 72
  Grade 5 event
Frequency of Grade 2, 3 or 4 AEs | Measured through Week 72
  Based on labs, signs/symptoms, diagnoses
Frequency of Grade 2, 3 or 4 AEs judged by the CMC to be related to DLM | Measured through Week 72
  Based on labs, signs/symptoms, diagnoses
Frequency of change in QTcF interval from baseline of greater than 60 ms | Measured through Week 72
  Based on ECG

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Garcia-Prats, MD, Study Chair — University of Stellenbosch; Ethel Weld, MD, Study Chair — Johns Hopkins University
Locations (5):
- Byramjee Jeejeebhoy Medical College (BJMC) CRS, Pune, Maharashtra, India
- South Africa (3):
  - Sizwe CRS, Johannesburg, Gauteng
  - PHRU Matlosana CRS, Klerksdorp, North West
  - Desmond Tutu TB Centre - Stellenbosch University (DTTC-SU) CRS, Cape Town, Western Cape
- Kilimanjaro Christian Medical Centre (KCMC), Moshi, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the International Maternal Pediatric Adolescent AIDS Clinical Trial (IMPAACT) Network by NIH.
Access Criteria: * With whom?
    * Researchers who provide a methodologically sound proposal for use of the data that is approved by the IMPAACT Network.
  * For what types of analyses?
    * To achieve aims in the proposal approved by the IMPAACT Network.
  * By what mechanism will data be made available?
    * Researchers may submit a request for access to data using the IMPAACT "Data Request" form at: https://www.impaactnetwork.org/resources/study-proposals.htm. Researchers of approved proposals will need to sign an IMPAACT Data Use Agreement before receiving the data.

REFERENCES:
- See also: Related Info — http://impaactnetwork.org/studies/IMPAACT2005.asp